CLINICAL TRIAL: NCT04341701
Title: Phenotype Identification Based on Multimodal MRI Analysis of Patients With Bronchial Obstructive Diseases
Acronym: PIMABOD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2018/37
Record Dates: First submitted 2020-04-02; First posted 2020-04-10 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Asthma Copd
Keywords: MRI; multimodal; phenotypes; lung; heart

STUDY DESIGN:
Intervention Model Description: diagnostic imaging pilot study, exploratory, prospective, multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD (Other): COPD according to GOLD 2019 but unrestricted to any level of bronchial reversibility established by the pulmonologist
  Interventions: Procedure: MRI
- Asthma (Other): asthma according to GINA 2019 but without any smoking restriction
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — The procedure to study lung and heart MRI, performed on a 1.5T magnet (Siemens), without any injection or inhalation of contrast agent

SUMMARY:
The hypothesis is that pulmonary and cardiac proton MRI allows phenotyping of patients with bronchial obstruction by cluster analysis based on quantitative multimodal imaging of bronchi, pulmonary vessels, pulmonary parenchyma, right and left ventricular function, myocardial fibrosis and pulmonary arterial pressure.

Such imaging will also offer the advantage of being non-irradiating and without contrast products, which will ultimately allow CT to be replaced by MRI in the follow-up of bronchial obstructive patients, thus avoiding the risks associated with repeated exposure to ionizing radiation.

DETAILED DESCRIPTION:
Bronchial obstructive diseases such as asthma and chronic obstructive pulmonary disease (COPD) are very common and represent a major public health problem. The distinction between these two diseases is sometimes difficult. In each of these diseases, several clinical phenotypes or biological endotypes have been defined. For example, frequent exacerbating patients and / or hypereosinophilic patients are present in both diseases. In the severe states, cardiovascular comorbidities are the most frequent comorbidities and alter the prognosis.

In these chronic obstructive patients, computed tomography (CT) allows a multimodal analysis of the bronchial wall, the lung parenchyma and pulmonary vessels. CT also allows a score analysis of coronary plaques. However, irradiation is significant and increases with repeated examinations. CT does not allow a comprehensive analysis of cardiac function, or an estimate of pulmonary artery pressure.

Magnetic Resonance Imaging (MRI) is a proton non-ionizing alternative to CT, in particular when using 3D ultra-short echo-time (UTE) sequences. These 3D-UTE sequences decrease the effects of magnetic susceptibility and provide morphological and morphometric information on bronchi and lung comparable to those obtained by CT. Moreover, dedicated sequences add functional information on bronchi. Heart MRI allows more analyses, such as right and left ventricular systolic functions, an indirect estimate of pulmonary arterial pressure and the amount of diffuse myocardial fibrosis.

Our project aims to identify morphological phenotypes through the pulmonary and heart MRI in patients with obstructive lung disease

.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged between 40 and 70 years.
* Having benefited under the current care of spirometry showing FEV / FVC pre-bronchodilation <0.70 at steady state (i.e., without exacerbation from at least 4 weeks).
* Having a diagnosis of asthma according to GINA 2019 without smoking restrictions or COPD according to GOLD 2019 but unrestricted to any level of bronchial reversibility to bronchodilator established by the pulmonologist.
* On stable cardiopulmonary medications for at least 4 weeks
* Having given his written informed consent.

Exclusion Criteria:

* Subject deprived of liberty by judicial or administrative decision.
* Major protected by law.
* Subject not affiliated to a social security scheme, whether or not the beneficiary of such a regime.
* Pregnant or breastfeeding women
* Inability to complete the Questionnaire SF-36 and SGQLQ.
* Subject in times of exclusion in relation to another protocol.
* History of pulmonary fibrosis, primary pulmonary hypertension and cystic fibrosis.
* History of lung resection (referred to oncological or volume reduction)
* History of cancer except skin cancer (squamous and Basal) under 5 years
* History of chest radiation
* Pacemaker carrier subject or implantable defibrillator, intraocular metallic foreign body, metal clip intracranial, heart valve prosthesis kind Starr-Edwards pre-6000, or biomedical insulin pump type device, Neurostimulator or cochlear implant, Metal patches.
* Subject claustrophobic or unable to stay elongate during 30 minutes.
* Subject with a waist circumference greater than 200 cm.
* Occurrence of an exacerbation between the FE and MRI
* Uninterpretable MRI

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Determine the number of the clusters | Day 30
  Number of the clusters will be defined using principal component analysis and dendrogram, based on the multimodal lung and heart MRI analysis
Determine the Quality of the clusters | Day 30
  Quality of the clusters will be defined using Dunn index and non-hierarchical analysis based on the multimodal lung and heart MRI analysis

SECONDARY OUTCOMES:
Assessment of age | Day 1
Assessment of sexe | Day 1
Assessment of tobacco consumption | Day 1
Assessment of disease duration | Day 1
Evaluation score of SF-36 questionnaire | Day 1
  Determine the quality of life. SF36: 36-Item Short Form health survey Minimum = 0 and maximum = 100 Higher score means better outcome
Evaluation with St Georges Quality of Life Questionnaire | Day 30
  Determine the quality of life. Minimum = 0 and maximum = 100 Higher score means worse outcome
Evaluation of comorbidities | Day 1
  The presence of various comorbidities will be checked in a yes/No manner :
  * rhinitis
  * sinusitis
  * nasal polyposis
  * gastroesophageal reflux
  * obstructive sleep apnea
  * depression
  * anxiety
  * allery
  * heart failure (Left or Right)
  * hypertension
  * myocardial infarction
  * stroke
  * arteriopathy
  * arythmia
  * diabetis
  * dyslipidaemia
  * obesity
  * denutrition
  * osteoporosis
Determine of Forced Expiratory Volume in one sec (FEV-1) during spirometry before and after bronchodilator | day 1
  Assessment of FEV-1/FVC during spirometry before and after bronchodilator
Determine of Forced Vital Capacity (FVC) during spirometry before and after bronchodilator | day 1
  Assessment of FEV-1/FVC during spirometry before and after bronchodilator
Determine of slow Vital Capacity (VC) during spirometry before and after bronchodilator | day 1
Determine of Total Lung Capacity (TLC) during spirometry before and after bronchodilator | day 1
Determine of Functional Residual Capacity (FRC) during spirometry before and after bronchodilator | day 1
Determine of Residual Volume (RV) during spirometry before and after bronchodilator | day 1
Determine of Carbon monoxide transfer capacity (TLCO) | day 1
Determine the value of blood heamoglobin | day 1
Determine the value of blood eosinophils | day 1
Determine the value of blood C-reactive protein | day 1
Determine the value of blood B-type natriuretic peptide | day 1
Determine the value of blood total IgE at | day 1
Determine the value of blood total IgE | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Patrick BERGER, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (6):
- France (6):
  - Centre hospitalier de la Côte Basque, Bayonne
  - Clinique Saint Augustin, Bordeaux
  - Centre Médical Toki Eder, Cambo-les-Bains
  - Hôpital Le Cluzeau - CHU de Limoges, Limoges
  - Centre de Pneumologie Bordeaux Rive droite, Lormont
  - Hôpital Haut-Lévêque - CHU de Bordeaux, Pessac

IPD SHARING:
Plan to Share IPD: No